

# The REST Trial

pRotective vEntilation with veno-venouS lung assisT in respiratory failure

| Protocol Number: | 15084DMcA-AS |
|---------------------|-----------------------------|
| | 16/SC/0089 (England, |
| Rec Number: | Wales and Northern Ireland) |
| | 16/SS/0048 (Scotland) |
| | NCT02654327 |
| Trial Registration: | |
| | ISRCTN 31262122 |

#### STATISTICAL ANALYSIS PLAN

Version 1.0 [Final] 16/12/19

**Contacts** 

### **Northern Ireland Clinical Trials Unit**

1st Floor Elliott Dynes The Royal Hospitals Grosvenor Rd Belfast BT12 6BA

**Tel:** +44 (0)28 96151447

Email: info@nictu.hscni.net

This document and all preceding versions will be stored in the Trial Master File for this trial

Doc No: ST06-RD01

Page **1** of **35** 

Danny McAuley: Chief Investigator

James McNamee: Clinical Lead

Clíona McDowell: Statistician

### Contents

| ABBRE\ | /IATIONS | . 3 |
|-------------|---------------------------------------------------------|-----|
| 1. | Background and Design | |
| 1.1 | Primary objective | |
| 1.2 | Secondary objectives | . 5 |
| 1.3 | Inclusion criteria | . 6 |
| 1.4 | Exclusion criteria | |
| 1.5 | Study Schematic Diagram | . 8 |
| 2. | Outcome measures | 9 |
| 2.1 | Primary outcome measure(s) | |
| 2.2 | Secondary outcome measures | . 9 |
| 2.3 | Exploratory Outcome Measures | .9 |
| 3. | Data | . 9 |
| 3.1 | CRF Forms and variables | |
| 3.2 | Management of datasets | 10 |
| 3.3 | Data completion schedule | 10 |
| 3.4 | Data verification | 13 |
| 3.5 | Data coding | 13 |
| 4. | Definition of terms | 13 |
| 5. | Sample Size Calculations | 14 |
| 6. | RANDOMISATION AND BLINDING | 15 |
| 6.1 | Randomisation | 15 |
| 6.2 | Blinding and Allocation Concealment | 16 |
| 7. | Analysis Principles | 16 |
| 7.1 | Subgroup analyses | |
| 8. | Analysis Details | |
| <b>8.</b> 1 | Recruitment and follow-up patterns | |
| 8.2 | CONSORT Flow Diagram | |
| | - | |
| 9. | Additional Information | |
| 9.1 | Trial Steering Committee (TSC) | |
| 9.2 | Data Monitoring and Ethics Committee (DMEC) | |
| 10. | Signatures of Approval | |
| | dix 1: P/F ratio reference table for inclusion criteria | |
| | dix 2: PEEP/FiO2 table | |
| Append | dix 3: Example Draft Summary Tables | 25 |

### **ABBREVIATIONS**

ABBREVIATION DEFINITION

ABG Arterial Blood Gas

AD8 Dementia Screening Interview

ADE Adverse Device Effect

AE Adverse Event

APACHE II Acute Physiology and Chronic Health Evaluation score

APRV Airway Pressure Release Ventilation
ARDS Acute Respiratory Distress Syndrome

CI Confidence Interval

CL Clinical Lead

CMP Case Mix Programme

CO<sub>2</sub> Carbon Dioxide

CPAP Continuous Positive Airway Pressure

CRF Case Report Form

DMEC Data Monitoring and Ethics Committee

DMP Data Management Plan

DNAR Do Not Attempt Resuscitation

ECCO<sub>2</sub>R Extracorporeal Carbon Dioxide Removal ECMO Extracorporeal Membrane Oxygenation

EQ-5D-5L EuroQoL-5 Dimension Questionnaire (5 level version)

FiO<sub>2</sub> Fraction of Inspired Oxygen

GP General Practitioner
HDU High Dependency Unit

HFOV High Frequency Oscillatory Ventilation

HRQoL Health Related Quality of Life

HSCIC Health and Social Care Information Centre

HTA Health Technology Assessment

ICNARC Intensive Care National Audit & Research Centre
ICH International Conference on Harmonisation

ICU Intensive Care Unit

MoCA-BLIND Montreal Cognitive Assessment/MoCA-Blind

NHS National Health Service

NICTU Northern Ireland Clinical Trials Unit
NIHR National Institute for Health Research

NMBD Neuromuscular Blocking Drugs

PaCO<sub>2</sub> Partial Pressure of Carbon Dioxide in arterial blood

PaO<sub>2</sub> Partial Pressure of Oxygen in arterial blood

PBW Predicted Body Weight

PEEP Positive End Expiratory Pressure

Doc No: ST06-RD01 Page **3** of **35**  P/F Ratio PaO<sub>2</sub>/FiO<sub>2</sub> ratio

PTSS 14 Post Traumatic Stress Syndrome Questionnaire

QoL Quality of Life RR Respiratory Rate

SADE Severe Adverse Device Effect

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SD Standard Deviation

SGRQ St George's Respiratory Questionnaire
SICSAG Scottish Intensive Care Society Audit Group

SOFA Sequential Organ Failure Assessment

SOP Standard Operating Procedures

TAPSE Tricuspid Annular Plane Systolic Excursion

TSC Trial Steering Committee

USADE Unanticipated Suspected Serious Adverse Device

Effect

VFDs Ventilator Free Days

Vt Tidal Volume

VV-ECCO<sub>2</sub>R Veno-venous Extracorporeal Carbon Dioxide Removal

Doc No: ST06-RD01

1. BACKGROUND AND DESIGN

The aim of this study proposes to deliver a multi-centre clinical trial to determine whether veno-

venous extracorporeal carbon dioxide removal (VV-ECCO<sub>2</sub>R) and lower tidal volume mechanical

ventilation improves outcomes and is cost-effective, in comparison with standard care in

patients who are mechanically ventilated for acute hypoxaemic respiratory failure.

Hypothesizing that in adult patients who require invasive mechanical ventilation for acute

hypoxaemic respiratory failure, VV-ECCO<sub>2</sub>R and lower tidal volume ventilation results in

reduced mortality.

This is a randomised, allocation concealed, controlled, open, pragmatic clinical and cost

effectiveness trial. The study objectives are as follows:

1.1 Primary objective

To determine whether VV-ECCO<sub>2</sub>R and lower tidal volume mechanical ventilation in patients

with acute hypoxaemic respiratory failure decreases mortality 90 days after randomisation.

1.2 Secondary objectives

In mechanically ventilated patients with acute hypoxaemic respiratory failure we want to

determine the effects of VV-ECCO<sub>2</sub>R on:

i. Tidal volumes

ii. Duration of mechanical ventilation

iii. Requirement for Extracorporeal Membrane Oxygenation (ECMO)

iv. Long-term mortality

v. Health Related Quality of Life

vi. Safety

vii. Cost-effectiveness in the NHS setting

viii. Long term respiratory morbidity

Patients will need to be assessed using the inclusion and exclusion criteria as set out below.

Eligibility to participate in the trial will be confirmed by a medically qualified person who is

Doc No: ST06-RD01

named on the Delegation Log. The medical care given to, and medical decisions made on behalf of subjects will be the responsibility of an appropriately qualified treating physician.

Two arterial blood gas samples (ABG) will be required but these will be collected as part of standard care. The P/F ratio table in appendix 1 can be used for reference.

Patients will be eligible to participate in the study if they fulfil the following criteria:

### 1.3 Inclusion criteria

- Invasive mechanical ventilation using PEEP ≥ 5cmH<sub>2</sub>O\*
- Acute and potentially reversible cause of acute respiratory failure as determined by the treating physician
- Within 48 hours of the onset of hypoxaemia as defined by PaO<sub>2</sub>/FiO<sub>2</sub> ≤ 20kPa\*\*

#### 1.4 Exclusion criteria

- Age < 16 years old</li>
- Intubated and mechanically ventilated via an endotracheal or tracheostomy tube ≥ 7
   days (168 hours) up to the time of randomisation
- Ability to maintain Vt to ≤ 3ml/kg PBW while maintaining pH ≥ 7.2 as determined by the treating physician\*
- Receiving, or decision to commence, ECMO in the next 24 hours.
- Mechanical ventilation using High Frequency Oscillatory Ventilation (HFOV) or Airway Pressure Release Ventilation (APRV)
- Untreated pulmonary embolism, pleural effusion or pneumothorax as the primary cause of acute respiratory failure.


<sup>\*</sup>Recommended on low tidal volume ventilation ≤ 6ml/kg PBW

<sup>\*\*</sup>Requires two ABG with a PaO2/FiO2  $\leq$  20kPa separated by at least 6 hours. 48 hour duration to consent begins at the time of 2nd ABG demonstrating PaO2/FiO2 ratio  $\leq$  20kPa. Site will then have a further 8 – 24 hours to randomise and administer the intervention. The onset of hypoxaemia is from time of intubation and invasive ventilation.(ABGs with PaO2/FiO2  $\geq$  20kPa are permitted between the two trial inclusion ABGs).

- Acute respiratory failure fully explained by left ventricular failure or fluid overload (May be determined by clinical assessment or echocardiography/cardiac output monitoring).
- Left ventricular failure requiring mechanical support
- Contra-indication to limited systemic anticoagulation with heparin
- Unable to obtain vascular access to a central vein (internal jugular or femoral vein)
- Inferior vena cava filter (if using femoral vein catheter)
- Consent declined
- Treatment withdrawal imminent within 24 hours
- Patients not expected to survive 90 days on basis of premorbid health status
- Do Not Attempt Resuscitation (DNAR) order (excluding advance directives) in place
- Severe chronic respiratory disease requiring domiciliary ventilation (except for sleep disordered breathing)
- Severe chronic liver disease (Child Pugh >11)
- Platelet count < 40,000 mm<sup>3</sup> (Prior to catheter insertion)
- Previously enrolled in the REST trial
- Prisoners

Full details of the background to the trial and its design are presented in the protocol.


<sup>\*</sup> This exclusion criterion relates to whether a Vt  $\leq$  3ml/kg PBW could be achieved without the need for ECCO<sub>2</sub>R. A tidal volume  $\leq$  3ml/kg is unlikely to be achievable in most clinical scenarios without ECCO<sub>2</sub>R as it is approaching dead space ventilation.

#### 1.5 **Study Schematic Diagram**

Figure 1: Study Schematic




### 2. OUTCOME MEASURES

### 2.1 Primary outcome measure(s)

All cause mortality 90 days after randomisation

### 2.2 Secondary outcome measures

- I. Tidal volume (ml/kg PBW) at day 2 and day 3 after randomisation
- II. Ventilator free days at 28 days after randomisation
- III. Duration of ventilation in survivors after randomisation at 28 days
- IV. Need for ECMO up to Day 7
- V. Mortality rate at 28 days, 6 months and 1 year after randomisation
- VI. Health Related Quality of Life (HRQoL) at 6 months and 1 year after randomisation
- VII. Adverse event rate
- VIII. Health & Social Care Service costs at 6 months and 1 year
  - IX. St George's Respiratory Questionnaire (SGRQ) at 1 year and need for home oxygen at 6 months and 1 year after randomisation
  - X. Post Traumatic Stress Syndrome Questionnaire (PTSS-14) at 1 year after randomisation
- XI. Montreal Cognitive Assessment (MoCA-BLIND) or AD8 Dementia Screening Interview (AD8) at 1 year after randomisation

### 2.3 Exploratory Outcome Measures

Right heart function as determined by echocardiography during 6ml/kg PBW and ≤3ml/kg PBW tidal volume ventilation (ECHO data will only be collected at a selected number of sites).

### 3. DATA

#### 3.1 CRF Forms and variables

Full details of the data to be collected and the timing of data collection are described in the trial protocol.

Doc No: ST06-RD01 Page **9** of **35**  A copy of the CRFs and questionnaires (e.g. Quality of Life (QoL) questionnaires) are presented in the Trial Master File.

### 3.2 Management of datasets

At the time of analysis:

The Data Manager in collaboration with the Study Statistician will extract data from MACRO following procedures as detailed in the SOP DM09 Database Closure/Lock and the corresponding study Data Management Plan (DMP).

### 3.3 Data completion schedule

### **Study Visits and Procedures**

Clinical data will be collected during trial participants stay in the ICU up to 28 days after randomisation. For routinely collected clinical data the NHS record will be the source document and for study specific clinical measurements the CRF will be the source document.

### Day 0 (baseline)

Day 0 is 24 hours prior to randomisation. If more than one value is available for this 24-hour period, the value closest but prior to the time of randomisation will be recorded. Day 0 (baseline) data collected will include but is not limited to:

- Patient demographics (date of birth, gender, measured height)
- ICNARC Case Mix Programme (CMP) number
- Scottish Intensive Care Society Audit Group (SICSAG) number
- Date/time of consent and randomisation
- Date and time of ICU admission
- Admission diagnostic category
- Assessment of functional status
- Presence of Acute Respiratory Distress Syndrome (ARDS) and aetiology
- Date/time of onset of mechanical ventilation
- The Acute Physiology and Chronic Health Evaluation score (APACHE II)


- PaO<sub>2</sub>/FiO<sub>2</sub> ratio (Qualifying PaO<sub>2</sub> /FiO<sub>2</sub> ratios including date/time)
- Date and time of worst PaO<sub>2</sub>/FiO<sub>2</sub> ratio
- Determinants of Sequential Organ Failure Assessment (SOFA) score
- Ventilation parameters including but not limited to: Mode of ventilation, minute volume, RR, mean airway pressure, plateau pressure, PEEP
- Arterial blood gas including but not limited to FiO<sub>2</sub>, PaO<sub>2</sub>, PaCO<sub>2</sub>, pH
- Date/time onset of ECCO<sub>2</sub>R therapy (from commencement of CO<sub>2</sub> removal)
- Use of adjunctive therapies including Neuromuscular Blocking Drugs (NMBD) and prone position
- Echocardiography parameters including but not limited to ventricular size and function and tricuspid annular plane systolic excursion (TAPSE)

### **Daily Data:**

Day 1 is from the time of randomisation to the end of that calendar day. If more than one value is available for this period, the value closest but after the time of randomisation will be recorded. All other daily measurements will be recorded and collected between 6-10am or as close to this time as possible, unless otherwise stated in the CRF. Daily data will be collected to day 7 and will include but is not limited to:

- Ventilation parameters including but not limited to: Mode of ventilation, minute volume, RR, mean airway pressure, plateau pressure, PEEP
- Arterial blood gas including but not limited to FiO<sub>2</sub>, PaO<sub>2</sub>, PaCO<sub>2</sub>, pH
- CO<sub>2</sub> removal rate while on ECCO<sub>2</sub>R therapy
- Commencement or transfer for ECMO following randomisation
- Use of adjunctive therapies including NMBD and prone positioning
- Blood product administration (blood, platelets, fresh frozen plasma, cryoprecipitate or other)
- Adverse events

### Day 1 and 2:

Echocardiography parameters including but not limited to ventricular size and function and TAPSE.


### **Day 3 and 7**

• Determinants of SOFA score

### 28 days:

Adverse Events

### 6 months:

- EuroQoL-5 Dimension Questionnaire (EQ-5D-5L) (Post or telephone)
- Patients use of health and social care resources collected by resource logs

#### 1 year:

- EQ-5D-5L (Post or telephone)
- Patients use of health and social care resources collected by resource logs
- SGRQ
- PTSS-14
- MoCA-Blind or AD8

The following data will also be collected

- Date of discontinuation of ECCO<sub>2</sub>R and reason
- Date of discontinuation of mechanical ventilation (unassisted breathing)
- Date of critical care discharge
- Date of hospital discharge
- Date of death

### **Follow Up Visits and Procedures**

HRQoL and Health and Social Care Service use will be assessed at 6 months and 1 year after randomisation. Patients will also be required to complete the SGRQ at 1 year.

The CTU will also collect mortality data at 1, 2 and 5 years post randomisation.


#### 3.4 Data verification

Study specific data validation checks will be implemented. The process of data validation ensuring the accuracy and quality of the data will be carried out according to SOP DM04 Data Validation and Discrepancy Management.

### 3.5 Data coding

The variable codings will be as specified on the CRF.

## 4. **DEFINITION OF TERMS**

| Term | Definition |
|---|---|
| Discharge from | First discharge to a medical ward in the hospital or another hospital; |
| critical care | a transfer between ICUs is not considered a discharge from critical |
| | care. |
| Hospital discharge | Hospital discharge is the first date that the patient is discharged to |
| | home/ community, a transfer between hospitals is not considered |
| | as a hospital discharge |
| Unassisted | Extubated with supplemental oxygen, or room air, or open T-tube |
| breathing i.e. no | breathing, or tracheostomy mask breathing, or CPAP $\leq$ 5 cm H <sub>2</sub> O |
| ventilatory support | without pressure support for a calendar day. Patients receiving |
| | pressure support via non-invasive ventilation will be defined as |
| | receiving ventilatory support (except for sleep disordered |
| | breathing). |
| VFDs to day 28 | The number of days from the time of initiating unassisted breathing |
| | to day 28 after randomisation, assuming survival for at least two |
| | consecutive calendar days after initiating unassisted breathing and |
| | continued unassisted breathing to day 28. If a patient returns to |
| | assisted breathing and subsequently achieves unassisted breathing |

Doc No: ST06-RD01 Page **13** of **35**  to day 28, VFDs will be counted from the end of the last period of assisted breathing to day 28. A period of assisted breathing lasting less than 24 hours and for the purpose of a surgical procedure will not count against the VFD calculation. If a patient was receiving assisted breathing at day 27 or dies prior to day 28, VFDs will be zero. Patients transferred to another hospital or other health care facility will be followed to day 28 to assess this endpoint.

Duration of ventilation

Counted from recruitment to the end of the last period of assisted breathing

### 5. SAMPLE SIZE CALCULATIONS

The required sample size is 1120 patients. With 90% power at a p value of 0.05 with a 3% dropout, 560 per group will be required to detect a 23% relative reduction (9% absolute reduction) in 90 day mortality, assuming a control group mortality of 41%. This sample size would also detect a 20% relative reduction (8% absolute reduction) at 80% power.

We have used two independent sources for the estimation of the all-cause mortality that was used to determine the sample size:

- 1. Data from the Intensive Care National Audit and Research Centre (ICNARC) case mix programme (CMP) for UK intensive care patients. The unpublished ICNARC data from the CMP for the year 2012 was compiled from 133,266 admissions from 203 adult critical care units in England, Wales and Northern Ireland. For patients with a  $PaO_2/FiO_2$  ratio < 20kPa the ICU mortality was 40.7% and the hospital mortality was 48.8%.
- 2. Data from the NIHR HTA funded OSCAR trial (30). This was a recent large randomised controlled trial on high frequency oscillatory ventilation (HFOV) in patients with respiratory failure. The 30-day mortality in the control group in the OSCAR trial was 41.1%. These patients received conventional ventilation with a tidal volume of 6-8ml/kg PBW and had an average PaO<sub>2</sub>/FiO<sub>2</sub> ratio of 15kPa.

Doc No: ST06-RD01 Page **14** of **35**  We have assumed 90-day control group mortality will be at least equivalent to 41%. We have

used the effect size of one of the few interventions to reduce mortality in patients with

hypoxaemic respiratory failure. The ARDSNet ARMA trial demonstrated a 9% absolute risk

reduction in patients with hypoxaemic respiratory failure secondary to ARDS with lung

protective ventilation. Our hypothesis is that we can extend the benefits of more protective

lung ventilation with the use of ECCO<sub>2</sub>R. Loss to follow up in UK critical care trials is low. We

know this is approximately 3% from previously published research as well as from the

experience of our team in managing large critical care trials in the UK.

An independent statistician (for the DMEC) will conduct an interim analysis for the primary

outcome measure (mortality) before the recruitment of 560 patients; (half the estimated

sample size), to ascertain whether the assumptions made in the sample size calculations are

correct.

6. RANDOMISATION AND BLINDING

6.1 Randomisation

Once consent has been obtained for the patient to participate in the study the patient will be

randomised to either ECCO<sub>2</sub>R with lower tidal volume mechanical ventilation or standard care.

Patients will be randomised via a central randomisation system and sites will be provided with

trial specific randomisation guidelines. Randomisation will be completed by an appropriately

trained and delegated member of the research team.

Randomisation will be stratified by recruitment centre.

Participants will be allocated to ECCO<sub>2</sub>R with lower tidal volume mechanical ventilation or

standard care on a 1:1 ratio. At the time of randomisation, each patient will be allocated a

unique Participant Study Number, which will be used throughout the study for participant

identification. An entry will be recorded in the patient medical notes noting enrolment into the

study.

Doc No: ST06-RD01

The research team will then ensure that the clinical team are informed which treatment this process has allocated. They will liaise with the clinical team as required to ensure that the allocated treatment is administered. If allocated VV-ECCO<sub>2</sub>R, this should ideally be commenced within 8 hours of randomisation.

### 6.2 Blinding and Allocation Concealment

Only the allocation of the intervention will be concealed; once assigned to the standard care or intervention group the interventions will be unblinded to the trial participant's representative (and to the participant on regaining capacity), research team, care providers, data analysts and outcome assessors. By the nature of the intervention it will not be possible to blind clinicians to whether a participant has been randomised to ECCO<sub>2</sub>R or standard care.

### 7. ANALYSIS PRINCIPLES

The primary analysis will be conducted on all outcome data obtained from all participants as randomised and regardless of protocol adherence, i.e. intention to treat analysis.

Standard approaches will be used to detect patterns in missing data. Baseline characteristics, follow-up measurements and safety data will be described using the appropriate descriptive summary measures depending on the scale of measurement.

For the primary outcome and other dichotomous outcomes, risk ratios and 95% confidence interval (CI) will be calculated. The primary outcome of 90 day mortality will be analysed using chi-square and a secondary analysis using logistic regression to adjust for age, SOFA score, Baseline  $PaO_2$  / $FiO_2$  and Baseline Plateau Pressure will also be carried out. The comparison of continuous outcomes between the two groups will be investigated using analysis of variance/analysis of covariance (if baseline measurements available), adjusting for other covariates where appropriate. Time-to-event outcomes will be analysed by survival methods and reported as hazard ratios with 95% CI. The intention-to-treat basis analysis will use a significance level of <0.05 for the primary outcome. Sensitivity analysis will be performed for the primary outcome excluding the first two intervention arm patients at each site in order to address potential learning effects. This would be explored further using a power curve model.

Doc No: ST06-RD01 Page **16** of **35**  Per protocol analysis will also be carried out for the secondary outcome of Tidal Volume at Days 2 and 3 i.e. including those who were on VV-ECCO<sub>2</sub>R on day 2 and 3 in the intervention arm. Estimates of effects/association and 95% CI will be reported for secondary and exploratory outcomes.

An independent statistician (for the DMEC) will conduct an interim analysis for the primary outcome measure before the recruitment of 560 patients. Using the chi-square statistic (mortality by treatment group), a p value less than 0.001 will be used according to the Haybittle-Peto stopping rule.

### 7.1 Subgroup analyses

Exploratory analyses will be reported using 99% confidence intervals. Logistic regression will be used with interaction terms (treatment group by subgroup) for the following subgroups:

- (i) Presence of ARDS prior to randomisation
- (ii) Baseline PaO<sub>2</sub> /FiO<sub>2</sub> ratio prior to randomisation (<50/50-99/100-150)
- (iii) Baseline Plateau Pressure prior to randomisation quartiles
- (iv) Volume of ECCO₂R participants at center (<10/>=10)
- (v) Vasopressor requirement prior to randomisation (yes/no)
- (vi) Baseline PaCO<sub>2</sub> prior to randomisation quartiles
- (vii) Baseline driving pressure prior to randomisation quartiles
- (viii) Baseline risk of death score (Apache II) quintiles prior to randomisation.

### 8. ANALYSIS DETAILS

The results of the analyses will be reported following the principles of the ICH E3 guidelines on the Structure and Content of Clinical Study Reports.

#### 8.1 Recruitment and follow-up patterns

- Recruitment by site
- Withdrawals by site
- Mortality 1, 2 and 5 years post randomisation





#### 8.3 Baseline Characteristics

- Age, mean (SD) by treatment arm
- Gender, no. (%) by treatment arm
- Dependency prior to hospital admission, no. (%) by treatment arm
- Height (cm), mean (SD) by treatment arm
- Predicted body weight (kg), mean (SD) by treatment arm
- Admission diagnostic category, no. (%) by treatment arm
- Presence of ARDS, no. (%)by treatment arm
- Aetiology of Ards, no. (%) by treatment arm
- APACHE II score, mean (SD) by treatment arm
- Arterial blood gas PaCO<sub>2</sub>, mean (SD) by treatment arm
- PaO<sub>2</sub>/FiO<sub>2</sub> ratio closest to but prior to randomisation, mean (SD) by treatment arm
- Second qualifying PaO<sub>2</sub>/FiO<sub>2</sub> ratio, mean (SD) by treatment arm
- Worst PaO<sub>2</sub>/FiO<sub>2</sub> ratio, mean (SD) by treatment arm
- Arterial pH, mean (SD) by treatment arm
- Total SOFA score, mean (SD) by treatment arm
- Mode of ventilation, no. (%) by treatment arm
- Use of Adjunctive therapies, no. (%) by treatment arm
- Mean airway pressure (cmH<sub>2</sub>O), mean (SD) by treatment arm
- PEEP (cmH<sub>2</sub>O), mean (SD) by treatment arm
- Plateau Pressure (cmH<sub>2</sub>O), mean (SD) by treatment arm
- Total Respiratory Rate (breaths/min), mean (SD) by treatment arm
- Minute Volume (L/min), mean (SD) by treatment arm
- Tidal Volume (ml/kg PBW), mean (SD) by treatment arm

### 8.4 Trial treatment

- Treatment allocation (Intervention), no. (%) commencing ECCO<sub>2</sub>R
- Adherence to protocol-specified intervention, no. (%) by treatment arm receiving
   ECCO<sub>2</sub>R for >48 hrs
- Duration of ECCO<sub>2</sub>R mean(SD) days


#### 8.5 Trial Outcomes

- All-cause mortality 90 days after randomisation, no (%) by treatment arm, Risk ratio 95%
- Tidal Volume (ml/kg PBW) at days 2 and 3 after randomisation, mean (SD) by treatment arm, difference in mean with 95% CI
- Ventilator free days at 28 days after randomisation, mean (SD) by treatment arm,
   difference in mean with 95% CI
- Ventilation duration in survivors after randomisation at 28 days, mean (SD) by treatment arm, difference in mean with 95% CI
- Need for ECMO up to day 7, no (%) by treatment arm, Risk ratio 95% CI
- Mortality rate at 28 days after randomisation, no (%) by treatment arm, Risk ratio 95%
- Mortality rate at 6 months after randomisation, no (%) by treatment arm, Risk ratio 95%
- Mortality rate at 1 year after randomisation, no (%) by treatment arm, Risk ratio 95% CI
- SGRQ at 1 year after randomisation, Symptoms score, Activity score, Impacts score and
   Total score mean (SD) by treatment arm, difference in mean with 95% CI
- Need for home oxygen at 6 months and 1 year after randomisation, no (%) by treatment arm, Risk ratio 95% CI
- Post Traumatic Stress Syndrome Questionnaire (PTSS-14) at 1 year after randomisation,
   mean (SD) by treatment arm, difference in mean with 95% CI
- Montreal Cognitive Assessment (MoCA-BLIND) or AD8 Dementia Screening Interview (AD8) at 1 year after randomisation, mean (SD) by treatment arm, difference in mean with 95% CI
- Right heart function as determined by echocardiography during 6ml/kg PBW and
  ≤3ml/kg PBW tidal volume ventilation. Echocardiography parameters including but not
  limited to ventricular size and function and TAPSE, mean (SD) by treatment arm,
  difference in mean with 95% CI


### 8.6 Toxicity/ Symptoms

• Adverse Event Rate, no. events (%) by treatment arm , no. patients (%) by treatment arm. Risk Ratio and 95% CI.

AEs of interest are as follows:

Device failure causing AE Haemolysis Bleeding

At cannula site

Other site

Infectious complications

Heparin induced thrombocytopenia

- Adverse Device Effect, no. events (%) by treatment arm, no. patients (%) by treatment arm. Risk Ratio and 95% CI.
- Serious Adverse Event, no. events (%) by treatment arm and System Organ Class, no.
   patients (%) by treatment arm. Risk Ratio and 95% CI.
- Serious Adverse Device Effect, no. events (%) by treatment arm and System Organ Class, no. patients (%) by treatment arm. Risk Ratio and 95% CI.
- Unanticipated Serious Adverse Device effect, no. events (%) by treatment arm and
   System Organ Class, no. patients (%) by treatment arm. Risk Ratio and 95% CI.

### 8.7 Health Economics

Details of the Health Economics analysis will be outlined in a separate Health Economics Analysis Plan.

## 9. ADDITIONAL INFORMATION

### 9.1 Trial Steering Committee (TSC)

The TSC will provide oversight with respect to the conduct of the study on behalf of the Funder and Sponsor. An independent chair will lead the TSC, with at least 75% independent membership. Membership and roles of the TSC will be listed in the TSC Charter. The TSC will incorporate a patient/public representative as well as the CI and CL.

Doc No: ST06-RD01 Page **21** of **35**  The TSC will meet at least annually and observers may be invited and be in attendance at TSC meetings, such as the Sponsor or Funder representatives or the Trial Manager to provide input on behalf of the CTU.

### 9.2 Data Monitoring and Ethics Committee (DMEC)

The independent DMEC will be comprised of at least 2 independent clinicians with experience in clinical trials, and an independent statistician. One of the independent clinicians will have experience in the regulatory aspects of clinical trials involving medical devices.

The role of the independent DMEC will be detailed in the DMEC charter but will include: monitoring the data and making recommendations to the TSC on whether there are any ethical or safety reasons why the trial should not continue; considering the need for any interim analysis; advising the TSC regarding the release of data and/or information; considering data emerging from other related studies. The independent DMEC will meet at least 6 monthly and additional meetings can be convened if the event of any safety concerns.

If funding is required above the level originally requested, the independent DMEC may be asked by the CI, TSC, Sponsor or Funder to provide advice and, where appropriate, information on the data gathered to date in a way that will not compromise the trial.


### 10. SIGNATURES OF APPROVAL

Date:

24th December 2019

Version:

1.0 Final

This document has completed a final review and is understood and approved by the following:

Danny McAuley

Chief Investigator Signature

Date dd/mm/yyyy

Cliona McDowell

Cliona McDowell

Cliona McDowell

Cliona McDowell

Study Statistician Signature

Date dd/mm/yyyy

Appendix 1: P/F ratio reference table for inclusion criteria

| FiO <sub>2</sub> | Maximum PaO2 if<br>P/F ratio ≤ 20kPa |
|------------------|--------------------------------------|
| 0.50 | 10.0 kPa |
| 0.55 | 11.0 kPa |
| 0.60 | 12.0 kPa |
| 0.65 | 13.0 kPa |
| 0.70 | 14.0 kPa |
| 0.75 | 15.0 kPa |
| 0.80 | 16.0 kPa |
| 0.85 | 17.0 kPa |
| 0.90 | 18.0 kPa |
| 0.95 | 19.0 kPa |
| 1.00 | 20.0 kPa |

### Appendix 2: PEEP/FiO2 table

| FiO <sub>2</sub> | 0.3 | 0.4 | 0.4 | 0.5 | 0.5 | 0.6 | 0.7 | 0.7 |
|------------------|-----|-----|-----|-----|-----|-----|-----|-----|
| PEEP | 5 | 5 | 8 | 8 | 10 | 10 | 10 | 12 |

| FiO <sub>2</sub> | 0.7 | 0.8 | 0.9 | 0.9 | 0.9 | 1.0 |
|------------------|-----|-----|-----|-----|-----|-------|
| PEEP | 14 | 14 | 14 | 16 | 18 | 18-24 |


### **APPENDIX 3: EXAMPLE DRAFT SUMMARY TABLES**

### Figure xxx. Recruitment by Site

### Figure xxx. Withdrawals by Site

Table x.x.x. Baseline Characteristics at trial entry

| Table A.A.A. Daseline Characteristics at that entry | ECCO₂R | Standard Care |
|---|---|---|
| | Intervention | n = (%) |
| | n = (%) | |
| Age (years) | | |
| Gender Male | | |
| Female | | |
| Dependency prior to hospital admission | | |
| Able to live without assistance in daily activities | | |
| Minor assistance with some daily activities | | |
| Major assistance with majority of/all daily activities | | |
| Total assistance with all daily activities | | |
| Height (cm) Measured length of patient (heel to crown) | | |
| Predicted body weight (kg) | | |
| Admission diagnostic category | | |
| Central Nervous System | | |
| Central Vascular System | | |
| Respiratory System | | |
| GIT Hepatology | | |
| Renal | | |
| Toxicology | | |
| Haematology | | |
| Orthopaedic | | |
| Sepsis | | |
| Other | | |
| Presence of ARDS | | |
| Aetiology of ARDS | | |

| | ECCO₂R | Standard Care |
|---|---|---|
| | Intervention | n = (%) |
| | n = (%) | |
| Smoke/toxin inhalation | | |
| Gastric content aspiration | | |
| Near drowning | | |
| Thoracic trauma | | |
| Pneumonia | | |
| Sepsis | | |
| Cardiopulmonary bypass | | |
| Pancreatitis | | |
| Non-thoracic trauma | | |
| Other | | |
| APACHE II score | | |
| Arterial blood gas PaCO <sub>2</sub> | | |
| PaO <sub>2</sub> :FiO <sub>2</sub> ratio | | |
| Worst PaO <sub>2</sub> /FiO <sub>2</sub> ratio | | |
| Second qualifying PaO <sub>2</sub> /FiO <sub>2</sub> ratio | | |
| Arterial pH | | |
| Total SOFA Score | | |
| Mode of Ventilation | | |
| Mandatory, no spontaneous additional breaths above | | |
| the fixed respiratory rate | | |
| Spontaneous, no back up mandatory breaths | | |
| Mixed, Mandatory and spontaneous breaths | | |
| Other | | |
| Use of Adjunctive therapies | | |
| NMBD | | |
| PP | | |
| INO | | |
| Other | | |
| Mean airway pressure (cmH <sub>2</sub> O) | | |
| PEEP (cmH <sub>2</sub> O) | | |
| Plateau Pressure (cmH₂O) | | |


| | ECCO <sub>2</sub> R Intervention n = (%) | Standard Care<br>n = (%) |
|---|---|---|
| Total Respiratory Rate (Breaths/min) | | |
| Minute volume (mL/min) | | |
| Tidal Volume (mls/kg PBW) | | |

Mean (SD) presented for continuous variables and no. (%) for all categorical variables.

### Table x.x.x. Treatment after Trial Entry

| | ECCO₂R | Standard Care |
|---|---|---|
| | Intervention | n = (%) |
| | n = (%) | |
| Treatment Allocation | | |
| Adherence to protocol-specified intervention | | |
| No. of days on ECCO₂R* | | |
| Reasons for ECCO <sub>2</sub> R Discontinuation | | |
| The patient's legal representative has requested | | |
| witdrawal from the study | | |
| There has been a safety concern about the therapy | | |
| such that withdrawal is mandated | | |
| <ul> <li>ECCO₂R therapy has been weaned</li> </ul> | | |
| <ul> <li>7 days post randomisation</li> </ul> | | |
| Escalation to ECMO has occurred | | |
| Discontinuation of active medical treatment has | | |
| occurred | | |
| The patient has died | | |
| Other | | |
| Protocol Deviations: | | |
| Eligibility | | |
| Treatment | | |
| Process | | |
| Other | | |

<sup>\*</sup>Mean (SD) no. of days on ECCO₂R


### **Table x.x.x Main Clinical Outcome variables**

| | ECCO₂R<br>Intervention n =<br>(%) | Standard Care<br>n = (%) | Difference<br>(95% CI) | p-value |
|---|---|---|---|---|
| Primary outcome; Mortality 90 days | | | | |
| post randomisation# | | | | |
| VFDs 28 days post randomisation | | | | |
| Ventilation duration post | | | | |
| randomisation | | | | |
| All | | | | |
| Survivors | | | | |
| Non-survivors | | | | |
| Need for ECMO to day 7 | | | | |
| Yes | | | | |
| No <sup>#</sup> | | | | |
| Mortality rate at 28 days post | | | | |
| randomisation <sup>#</sup> | | | | |
| Mortality rate at 6 months post | | | | |
| randomisation <sup>#</sup> | | | | |
| Mortality rate at 1 year post | | | | |
| randomisation <sup>#</sup> | | | | |
| SGRQ | | | | |
| Symptoms Score | | | | |
| Activity Score | | | | |
| <ul> <li>Impacts Score</li> </ul> | | | | |
| Total Score | | | | |
| Need for home oxygen at 1 year post | | | | |
| randomisation# | | | | |
| PTSS-14 Score | | | | |
| MoCA-Blind | | | | |
| AD8 Dementia Screening | | | | |

Mean (SD) presented for treatment arms

### Figure x.x.x. Kaplan Meier Curve

Time to death and no. of deaths on x-axis


<sup>\*</sup>No. (%) for treatment arms and Risk Ratio and 95% CI presented

Table x.x.x. Tidal Volume after Randomisation

| | ECCO₂R<br>Intervention<br>n = (%) | Standard Care<br>n = (%) | Mean Difference<br>(95% CI) |
|---|---|---|---|
| Tidal volume ml/kg PBW | | | |
| Day 2 | | | |
| Day 3 | | | |
| Day 4 | | | |
| Day 5 | | | |
| Day 6 | | | |
| Day 7 | | | |
| Tidal volume ml/kg PBW* | | | |
| Day 2 | | | |
| Day 3 | | | |

Mean (SD) and Min/Max presented for TV and no. (total % out of 40) for recruitment rate.


<sup>\*</sup>Per protocol population i.e. those who were on VV-ECCO<sub>2</sub>R on day 2 and 3 in the intervention arm

Table x.x.x. Safety by Treatment Group

| | | Number of events | | | Number of patients | | | |
|---|---|---|---|---|---|---|---|---|
| | | Total<br>n | Intervention<br>ECCO <sub>2</sub> R<br>n (%) | Standard Care<br>n (%) | Total<br>n (%) | Intervention<br>ECCO <sub>2</sub> R<br>n (%) | Standard<br>Care<br>n (%) | RR(95%CI) |
| AEs, SAEs, ADE,<br>SADE, USADE | Total SAEs | | | | | | | |
| | Related to study device | | | | | | | |
| | Related to study device and unanticipated | | | | | | | |
| | Total AEs | | | | | | | |
| | Related to study device | | | | | | | |
| SAEs | Cardiac Disorders | | | | | | | |
| | Hepatobiliary disorders | | | | | | | |
| | Respiratory, thoracic and mediastinal disorders | | | | | | | |
| | etc | | | | | | | |
| AEs | Device failure causing AE | | | | | | | |
| | Haemolysis | | | | | | | |
| | Bleeding at cannula site | | | | | | | |
| | Bleeding at other site | | | | | | | |
| | Infectious complications | | | | | | | |
| | Heparin induced thrombocytopenia | | | | | | | |
| Adverse Device effect | | | | | | | | |
| Serious Adverse<br>Device effect | | | | | | | | |

### The REST Trial STATISTICAL PLAN (Final version 1.0, 16/12/19)

| Unanticipated |
|-----------------|
| Serious Adverse |
| Device effect |

For no. of events %s are calculated within total SAEs, AEs, ADEs and SADEs respectively within treatment arm.


Table xxx. Follow-up Questionnaires at 1 year

| | ECCO₂R<br>Intervention n<br>= (%) | Standard Care<br>n = (%) | Difference<br>(95% CI) |
|---|---|---|---|
| Saint Georges | | | |
| Questionnaire | | | |
| PTSS-14 | | | |
| MoCA | | | |
| AD8 | | | |

### Figure x.x.x. Subgroup Analyses

### OR and 99% CI will be presented graphically alongside the n(%) for interaction terms for the following pre-specified subgroups

| | Treatment Group | | |
|---|---|---|---|
| | Intervention ECCO <sub>2</sub> R | Standard Care | Difference<br>(99% CI) |
| Presence of ARDS prior to randomisation | | | |
| Yes | | | |
| No | | | |
| Baseline PaO <sub>2</sub> /FiO <sub>2</sub> ratio prior to randomisation | | | |
| <50 | | | |
| 50-99 | | | |
| 100-150 | | | |
| Baseline Plateau Pressure prior to randomisation | | | |
| Quartile 1 | | | |
| Quartile 2 | | | |
| Quartile 3 | | | |
| Quartile 4 | | | |
| Volume of ECCO₂R participants at center | | | |
| <10 cases | | | |
| >=10 cases | | | |


### The REST Trial STATISTICAL PLAN (Final version 1.0, 16/12/19)

| | Treatment Group | | |
|---|---|---|---|
| | Intervention ECCO <sub>2</sub> R | Standard Care | Difference<br>(99% CI) |
| Vasopressor requirement prior to randomisation | | | |
| Yes | | | |
| No | | | |
| Baseline PaCO <sub>2</sub> prior to randomisation | | | |
| Quartile 1 | | | |
| Quartile 2 | | | |
| Quartile 3 | | | |
| Quartile 4 | | | |
| Duration of Carbon Dioxide (CO <sub>2</sub> ) removal | | | |
| Quartile 1 | | | |
| Quartile 2 | | | |
| Quartile 3 | | | |
| Quartile 4 | | | |
| Baseline driving pressure prior to randomisation | | | |
| Quartile 1 | | | |
| Quartile 2 | | | |
| Quartile 3 | | | |
| Quartile 4 | | | |
| Baseline risk of death score (Apache II) quintiles prior to | | | |
| randomisation | | | |
| Quintile 1 | | | |
| Quintile 2 | | | |
| Quintile 3 | | | |
| Quintile 4 | | | |
| Quintile 5 | | | |

### **Table x.x.x. Exploratory Outcome Measures**

| | Treatment Group | | |
|---|---|---|---|
| | Intervention ECCO₂R | Standard Care | Difference<br>(99% CI) |
| Baseline / Day 0: | | | |
| <ul> <li>Tricuspid annular plane systolic excursion (TAPSE) measured in cm</li> <li>Right ventricular strain (RVS) measured in percentage</li> <li>Right ventricle fractional area of change (FAC) measured in percentage</li> <li>Right ventricle end diastolic area to Left ventricle end diastolic ratio (EDA ratio) measure as a ratio (e.g. 0.6)</li> <li>Left ventricular end diastolic diameter measured in cm</li> <li>Left ventricle function measured in percentage</li> </ul> | | | |
| Day 1 or 2: | | | |
| <ul> <li>TAPSE measured in cm</li> <li>RVS measured in percentage</li> <li>Right Ventricle FAC measured in percentage</li> <li>Right ventricle EDA ratio</li> <li>Left ventricle end diastolic diameter measured in cm</li> <li>Left ventricle function measured in percentage</li> </ul> | | | |
